CLINICAL TRIAL: NCT01551784
Title: An Observational Study of Statin Treatment Induced HDL Changes - Effect on Cardiovascular Disease
Brief Title: An Observational Study of Statin Treatment Induced HDL Changes
Acronym: SIRIUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CSE-CRE-2011/1
Record Dates: First submitted 2012-03-05; First posted 2012-03-13 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Cardiovascular Disease
Keywords: Statin treatment; Cardiovascular disease; Statin treatment induced HDL changes and the effect on cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Cholesterol values (HDL-C, LDL-C, TC)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The aim with this study is to investigate the effect of statin induced changes in HDL-C on all cause mortality and CVD with adjustment for changes in other blood lipids and clinical parameters in Sweden, UK and the Netherlands.

DETAILED DESCRIPTION:
An observational study of statin treatment induced HDL changes - effect on cardiovascular disease

ELIGIBILITY:
Inclusion Criteria:

* Started treatment with statins within the observation period (2004-2010)
* The patient must have valid baseline and follow-up measurements for HDL-C and LDL-C.

Exclusion Criteria:

* Malignancy Alcohol abuse/alcohol dependence

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received a first prescription of a statin (ATC code C10AA) between 1st of January 2004 and 31st of December 2010. Swedish data will be extracted from medical records and national registers and for UK and the Netherlands from central registers.
Sampling Method: Non-Probability Sample
Enrollment: 120000 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Time to first occurrence of hospitalization for acute myocardial infarction, unstable angina pectoris or ischemic stroke related to changes in HDL-C | 1st of January 2004 to 31st December 2010

SECONDARY OUTCOMES:
The effect of statin induced changes in HDL-C (per mmol/L) on a composite endpoint including unstable angina pectoris, myocardial infarction, ischemic stroke and all cause mortality. | 1st of January 2004 to 31st December 2010
Time to first occurence of hospitalization for acute myocardial infarction, unstable angina pectoris or ischemic stroke and ischemic heart disease mortality related to changes in HDL-C. | 1st of January 2004 to 31st December 2010
The relationships between acquired HDL levels after statin treatment on the primary endpoint and the effect of HDL increase on the primary endpoint for different levels of baseline HDL | 1st of January 2004 to 31st December 2010
Potential interactions between baseline HDL and HDL increase and other factors like age, gender, treatment and co-morbidity on the primary endpoint | 1st of January 2004 to 31st December 2010
The health economic consequences of increasing HDL-C with statin treatment | 1st of January 2004 to 31st December 2010

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Johansson, MD, PROFESSOR, Principal Investigator — Department of Public Health and Caring Sciences, Family Medicine and Clinical Epidemiology Uppsala University 751 22 Uppsala Sweden; Ron Herings, DR, ASSOC PROF, Principal Investigator — Pharmo Institute for Drug Outcomes Research3508 AE UtrechtThe Netherlands